CLINICAL TRIAL: NCT05270707
Title: HyperArc Registry Study
Status: Completed | Type: Observational
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Other Study IDs: VAR-2019-01
Record Dates: First submitted 2022-02-14; First posted 2022-03-08 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Brain Metastases; CNS Neoplasm; CNS Disorder, Intracranial
Keywords: Stereotactic Radiosurgery
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Brain Diseases | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Radiation: Stereotactic radiosurgery — HyperArc is a radiotherapy treatment with a structured workflow to plan and deliver stereotactic radiosurgery (SRS).
  Other Names: HyperArc SRS

SUMMARY:
The HyperArc registry is designed to collect data from which the efficacy of the HyperArc procedure can be assessed and compared to alternative treatments.

DETAILED DESCRIPTION:
A significant percentage of newly diagnosed cancer patients will develop brain metastases. For many of these patients, stereotactic radiosurgery (SRS) is recommended as a primary treatment option. Concerns about complexity, patient safety, cost, and human resources can make SRS challenging. HyperArc radiotherapy addresses these challenges by introducing key technology and workflow elements to streamline multi-leaf collimator-based, non-coplanar SRS. HyperArc is designed to deliver SRS treatments from the TrueBeam linear accelerator platform. The HyperArc registry is designed to collect data from which the efficacy of the HyperArc procedure can be assessed and compared to alternative treatments.

ELIGIBILITY:
Inclusion Criteria:

* Received or scheduled to receive treatment using the HyperArc treatment method
* Age of legal adult according to local law
* Signed informed consent form, or, informed consent waived by the local ethics board/institutional review board

Exclusion Criteria:

* None, apart from not meeting Inclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient scheduled to be treated using the HyperArc method will be invited to participate, provided they meet other eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 968 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Survival | follow until death, on average approximately 2 years
  Survival

SECONDARY OUTCOMES:
Local tumor control | follow until death, on average approximately 2 years
  Response of treated tumors
HyperArc Patterns of Care | Limited to course of treatment: up to 4 weeks
  Dosimetry information for clinically delivered HyperArc treatments

CONTACTS AND LOCATIONS:
Locations (7):
- University of Alabama, Birmingham, Alabama, United States
- Australia (4):
  - Icon Cancer Centre Canberra, Bruce, Australian Capital Territory
  - Icon Cancer Centre Greenslopes, Greenslopes, Queensland
  - Icon Cancer Centre Maroochydore, Maroochydore, Queensland
  - Icon Cancer Centre Gold Coast Private, Southport, Queensland
- University Hospital Leuven, Leuven, Belgium
- L'IRCCS Ospedale Sacro Cuore - Don Calabria, Negrar, Valpolicella, Italy

IPD SHARING:
Plan to Share IPD: No